CLINICAL TRIAL: NCT04526392
Title: Pubertal Evolutionary Profile of Children Monitored for Fetal Ovarian Cyst
Acronym: KOF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0497
Record Dates: First submitted 2020-07-29; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Fetal Ovarian Cyst
Keywords: child; puberty
MeSH Terms: conditions — Neonatal ovarian cyst | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Patients will choose how they wish to complete the Pubertal Course Questionnaire: electronically (web link), on paper, by telephone, or face-to-face at a follow-up consultation.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Pubertal course questionnaire

SUMMARY:
This study is based on pubertal surveillance of fetal ovarian cysts (KOF). Fetal ovarian cysts (KOF) detected during fetal ultrasound examinations occur during the 3rd trimester of pregnancy and are of unknown cause.

DETAILED DESCRIPTION:
These cysts are functional in the vast majority of cases and are therefore likely to disappear spontaneously, but they may become complicated before regressing. Apart from complication, the natural evolution of these cysts, which are said to be "simple" because they are liquid on ultrasound, is towards regression in the first months of neo-natal life.

Surveillance during the 1st year of life showed that simple cysts regressed during the 1st trimester. In the case of complicated cysts, oophorectomy was necessary in 9 cases. In the 1-year follow-up, the ovarian recovery rate was significantly different depending on the appearance of the cyst (p<0.0001); 60 ovaries out of 89 homolateral to the cyst were follicular, of which 48/49 (98%) were carriers of fluid cysts and 12/40 (30%) were initially heterogeneous. The origin of these cysts is unknown, the ovary is again physiologically stimulated during the onset of puberty. No series in the literature gives the long-term ovarian prognosis for these patients. We wish to evaluate the pubertal evolutionary profile of patients followed at the University Hospital for KOF. The data collected concerning puberty (age of menses) will be examined in relation to the age of menses in the siblings and in the mother, as well as to the data in the literature on the age of the first menses in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 8 years of age at the time of inclusion.
* Patients being followed for fetal ovarian cyst.
* Minor patients of whom at least one of the two holders of parental authority has given his or her non-opposition.
* Patients covered by a social security scheme.

Exclusion Criteria:

* Patients less than 8 years of age at the time of inclusion
* Ovarian cysts outside the neonatal period
* Refusal to participate.
* Opposition to disclosure of neonatal data.
* Pregnant or nursing patient.

Ages: 8 Years to 18 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Young girls who have to answer a questionnaire on their pubertal development. Estimated duration of data collection by questionnaire for one participant: 30 minutes maximum.
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Age of onset of first menstruation | Day 1
  Age of onset of first menstruation defined with one decimal place (year and month).

SECONDARY OUTCOMES:
Average age of maternal and sister rules | Day 1
  Average age of maternal and sister menstruation.
Ovarian volumes | Day 1
  Homo and contralateral ovarian volumes at the cyst.
Presence or not of follicles | Day 1
  Presence or not of follicles on both ovaries.
first menstruation description - age of breast onset | Day 1
  Age of breast onset
first menstruation description - cycle length | Day 1
  cycle length in the last three months
first menstruation description - cycle disorder | Day 1
  rate of patients with cycle disorder
first menstruation description dysmenorrhoea. | Day 1
  dysmenorrhoea.
first menstruation description menorrhagia | Day 1
  menorrhagia
percentage of hyperandrogenism | Day 1
  Percentage of girls with clinical signs of hyperandrogenism or elevated testosterone levels.
Hormonal levels - AMH | Day 1
  AMH levels
Hormonal levels - LH | Day 1
  Luteinizing hormone (LH) levels
Hormonal levels - FSH | Day 1
  follicle stimulating hormone (FSH) levels
Hormonal levels - estradiol | Day 1
  estradiol levels
rate of ovarian cyst recurrence | Day 1
  Ovarian cyst recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PIENKOWSKI, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No